CLINICAL TRIAL: NCT02500771
Title: Feasibility Testing and Pilot Study of V-MOTIVE Protocol Software Version 1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Experiad LLC (Industry)
Collaborators: northwest behavioral associates (Unknown)
Responsible Party: Principal Investigator, Rex Jakobovits, President, Experiad LLC
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VMOTIVE-1
Record Dates: First submitted 2015-07-09; First posted 2015-07-17 (Estimated); Last update posted 2015-07-17 (Estimated); Status verified 2015-07

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- children and tutors using V-Motive (Experimental): The following intervention will be administered:
  ABA therapy enhanced with V-Motive software
  Tutors treating children with Applied Behavioral Analysis therapy will use the V-Motive software to enhance therapy sessions. Children will receive therapy as usual, but half of their current behavioral programs (skills/goals) will have been selected for enhanced prompting through video modeling.
  Interventions: Behavioral: ABA therapy enhanced with V-Motive software

INTERVENTIONS:
Behavioral: ABA therapy enhanced with V-Motive software — Tutors will use the V-Motive software to enhance their delivery of Applied Behavioral Analysis therapy.

SUMMARY:
This is a project to be funded by a Fast-Track Small Business Innovative Research to build and test the feasibility of a new software prototype called V-Motive which will facilitate the combination of two proven autism behavioral interventions: Applied Behavior Analysis therapy (ABA) and Video Modeling (VM). The investigators will conduct a Phase I feasibility analysis and Phase II pilot study of the V-Motive Prototype by observing a community therapy providers' use of the prototype in a therapy setting. Investigators will observe the users and record the success or failure of the performance of key functions of the software. Investigators will also administer surveys. The study will answer research questions about V-Motive's ability to perform its intended function: allowing interventionists to feasibly leverage video modeling within ABA therapy with a minimal amount of overhead and labor.

DETAILED DESCRIPTION:
Investigators will conduct a within-subject pilot study of 6 tutors and 6 children to answer research questions about V-Motive's ability to perform its intended function. The goal is to evaluate the feasibility, usability, and the potential of V-Motive to deliver comprehensive, individualized video modeling that is integrated with a child's program. Investigators will also use descriptive statistics to provide preliminary insight into the potential impact of the system on a child's performance in their ABA therapy. However, these data are NOT intended to show cause or to show effectiveness. The study will answer the following questions: 1) 3) Can V-Motive be feasibly used during ABA therapy to positively impact a child's performance within 4 weeks? 2) How laborious is it to construct a fully-indexed video repository from therapy footage using V-Motive? 3) How accurate is the system in suggesting and cueing up appropriate video for playback on demand?

ELIGIBILITY:
Inclusion Criteria:

* Children between 4 and 10 years old
* Clinical diagnosis of Autism Spectrum Disorder
* Currently receiving Applied Behavioral Analysis therapy
* Must be developmentally capable of basic imitation behavior

Exclusion Criteria:

- none

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2017-06; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility of V-Motive software's ability to positively impact a child's performance within 4 weeks | 4-week trial starting in 2020
  The following pilot feasibility measures will be captured for each tutor/child pair: 1) Usage: the total number of times the tutor chooses to use VM (an indicator that the tutor found it useful); 2) Overall Trial Success Rate: the percent of trials that were successful (e.g. recorded as a "pass") in programs with and without VM; 3) Mastery: the trials to criteria and the total number of targets mastered with and without VM; 4) Behavior Impact: the number of tantrums and other tracked behaviors occurring with and without VM (tracked by tutor using Abacus behavior tracker).

SECONDARY OUTCOMES:
Amount of time required to construct a fully-indexed video repository from therapy footage using V-Motive | 4-week trial starting in 2020
  Researchers will measure the time it takes to construct the video repository for each tutor (time spent setting up camera, initializing the upload process, etc).
Accuracy of V-Motive software in suggesting and cueing up appropriate video for playback on demand | 4-week trial starting in 2020
  The system will automatically capture the number of times a tutor adjusts the video for playback, number of times a video is rewound or fast-forwarded to obtain the appropriate start time, and the amount of time spent seeking before the video is cued up for playback to the child. For precision determination, actual start times will be obtained by manually reviewing the video of selected trials, and user seek times will be automatically tracked by the system.

CONTACTS AND LOCATIONS:
Overall Officials: Rex Jakobovits, Principal Investigator — Experiad LLC
Locations (1):
- Northwest Behavioral Associates, Bellevue, Washington, United States